CLINICAL TRIAL: NCT04884165
Title: Remote Monitoring to Improve Low Adherence in Non-invasive Ventilation: READ-NIV Trial
Brief Title: Remote Monitoring to Improve Low Adherence in Non-invasive Ventilation
Acronym: READ-NIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: READ-NIV 15-11-2020 V1.0; 270108 (Other: IRAS)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hypercapnic Respiratory Failure; Sleep Disordered Breathing; COPD; Obesity Hypoventilation Syndrome (OHS)
Keywords: Non-invasive ventilation; Home mechanical ventilation; Remote monitoring; Adherence; Compliance
MeSH Terms: conditions — Respiratory Insufficiency; Sleep Apnea Syndromes; Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Patient Compliance | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, parallel group controlled, unblinded clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Remote monitoring using SRETT (CE marked device) + home mechanical ventilation (non-invasive ventilation, NIV) and usual care.
  Interventions: Device: Remote monitoring of home mechanical ventilation (NIV) using SRETT
- Control (Active Comparator): Home mechanical ventilation (non-invasive ventilation, NIV) with usual care.
  Interventions: Other: Home mechanical ventilation (NIV) without remote monitoring

INTERVENTIONS:
Device: Remote monitoring of home mechanical ventilation (NIV) using SRETT — Patients will use the SRETT device attached to their home ventilator.
  Arms: Intervention
Other: Home mechanical ventilation (NIV) without remote monitoring — Usual care
  Arms: Control

SUMMARY:
Patients are invited to participate in a trial to test a new way to optimise long-term use of non-invasive ventilation using remote monitoring. Breathing difficulties during sleep are frequently treated using home mechanical ventilation, also called non-invasive ventilation (NIV). Breathing difficulties during sleep affect many patients with conditions such as chronic pulmonary obstructive disease (COPD), neuromuscular conditions and obesity hypoventilation syndrome. Left untreated they can cause breathlessness, headaches, sleepiness and lead to hospitalisations and other severe adverse health outcomes.

The best available treatment for chronic types of sleep-disordered breathing is NIV. However, not every patient eligible tolerates this treatment because it requires patients to sleep with a nasal or full-face mask that is connected with a tube to a machine. Although NIV is recommended by the National Institute for Health and Clinical Excellence (NICE), many patients who should be on NIV use the treatment insufficiently within months.

Using remote monitoring to identify problems with treatment adherence early on may help to identify clinical problems, troubleshoot user- or device-dependent problems, avoid delays in treatment and safe healthcare resources in the long-term.

The investigators invite patients who use NIV to participate in this trial when they have difficulties with the treatment (NIV). This study will evaluate compliance and efficacy of a remote monitoring device (T4P device, SRETT, Paris/France) that will be connected to the standard NIV machine to remotely monitor usage. Patients will be randomly assigned to the remote monitoring using NIV for three months at home, or to usual care which is NIV without this monitoring. The primary outcome measure of this study is the improvement in adherence and compliance, as indicated by the average usage of NIV, as well as symptom scores to assess treatment effects.

DETAILED DESCRIPTION:
Participant Selection

Patients established on NIV for >3months will be recruited in this trial. The sample size calculation of n=32 patients is based on previous in-house data (Ishak A et al, Respirology 2019 in press) to detect a difference in the treatment arms with a Power of >80% and an alpha of 5% using the improvement adherence as an outcome parameter.

Criteria and procedures for subject withdrawal or discontinuation.

Sample size estimation assumed 15-20% of patients would not provide end of study information that could be evaluated. If this rate is observed, data for some patients will be only partially observed. For patients who withdraw or drop out before the end of the study, the "no change assumption" will be used to impute the missing subsequent values. This may introduce a bias if the main reason for drop-out was deterioration. To examine this possibility, sensitivity analysis will be performed to assess the primary efficacy outcome using different imputation methods including "best-case scenario" and "worst- case scenario" possible scores for the missing data. A second per protocol analysis, including only those subjects with complete follow-up data will also be performed.

Subject Enrolment

Patients on NIV will be recruited from the Lane Fox Unit at Guy's & St Thomas' NHS Foundation Trust where they are assessed in clinics. The Lane Fox Unit runs daily outpatient clinics at the St Thomas' site. Currently, the Lane Fox Unit cares for >2,000 patients on home non-invasive ventilation.

The direct care team will approach patients after consultation with the Consultant and hand out a Patient Information Sheet to discuss the study with potential participants. Informed written consent will be taken after sufficient time to allow for information and questioning. Patients will then be offered a clinic date to come to hospital. If the patient fulfills all inclusion and no exclusion criteria, follow up will be booked at 6- weeks (phone call) and at 12-weeks (clinic appointment) following randomisation.

Procedures Informed Consent

A member of the direct clinical care team (Good Clinical Practice, GCP-trained) will take informed consent once the patients have had the opportunity to read and discuss the Patient Information Sheet with sufficient time. It will be clearly stated that the participant is free to withdraw from the study at any time without this affecting any future care and with no obligation to give the reason for withdrawal.

Following sufficient time and the opportunity to question the (Co-)investigator or other independent parties to decide whether they will participate in the study written informed consent will then be obtained. A copy of the signed informed consent will be given to the participants. The original signed form will be kept at the study site and a copy will be inserted in the medical notes.

Screening and Eligibility Assessment

Patients with sleep-disordered breathing and the need for non-invasive ventilation will be recruited from the Lane Fox Unit where they are assessed in the NIV clinics. The Lane Fox Unit runs daily outpatient clinics at the St Thomas' site. Currently, the Lane Fox Unit cares for >2,000 patients on home non-invasive ventilation.

The direct care team will approach patients after consultation with the Consultant and hand out a Patient Information Sheet to discuss the study with them. Informed written consent will be taken after sufficient time to allow for information and questioning. Patients will then be offered a date to come to hospital within four weeks for the baseline. If the patient fulfills all inclusion and no exclusion criteria, follow up will be booked at 6-weeks (phone call) and at 12-weeks (clinic appointment) following randomisation.

Baseline Assessments

The initial assessment will include an outpatient clinic appointment. Patients will be assessed using the following parameters:

1. Demographics i. Age ii. Gender iii. Height, Weight, Body-Mass-Index (BMI) iv. Neck circumference v. Waist, Hip, W:H ratio vi. Mallampati and Friedman Score vii. Basic lung function (spirometry: FEV1, FVC) viii. Blood pressure and heart rate ix. Medication use x. GP appointments/A&E contacts/hospitalisations (previous 3months)
2. Upper Airway i. Mallampati and Friedman score
3. Blood tests i. Arterial or earlobe blood gas analysis (including pH, pO2, pCO2, HCO3-)
4. Previous sleep study parameters, as measured when NIV was set up i. AHI/4%ODI ii. average SpO2 (%) iii. Total recording time iv. Diagnosis
5. Symptom and Quality of Life scores i. Epworth Sleepiness Scale (ESS) ii. Stanford Sleepiness Scale (SSS) iii. European Quality of Life tool (EQ-5D) iv. Hospital Anxiety and Depression Scale (HADS) v. Severe Respiratory Insufficiency questionnaire (SRI)
6. NIV adherence i. total hours used ii. average usage per night (hours) iii. total nights used

Randomisation

Randomisation and Home Treatment Following the baseline assessment, if eligible, patients will be randomized into active treatment (remote monitoring of NIV) or usual care (NIV). The active treatment will be remote monitoring at night while using NIV while the usual care group will receive ongoing NIV therapy without remote monitoring.

Randomisation will involve assigning a unique patient number in sequential, ascending chronological order (matched cases). This number will be a two-digit number prefixed by "R" (e.g. R01, R02 etc) and will be used to identify the treatment the patient was randomised to. Treatment assignment will be determined according to a computer generated randomisation list.

Subsequent assessments

Weekly Review of Online Data In the intervention group, the investigators will review the usage data weekly and, if it is found that the average usage for 3 subsequent nights is below 4 hours/night and/or the leak is >50L/min then the patient will be called to discuss any problems.

6-Week Telephone Contacts

All patients will receive a 6-week phone call to encourage NIV usage and discuss problems with the treatment. Patients will be asked about comfort and adverse events. The following parameters will be assessed:

i. Epworth Sleepiness Scale (ESS) ii. Stanford Sleepiness Scale (SSS) iii. subjective NIV usage (hours)

At this stage, the patients will be educated on the device/NIV again and encouraged to continue with the usage.

Follow up at 12-weeks

At 12-week follow up the patients will be invited to attend outpatient clinics at the Lane Fox Unit. The assessment will repeat the following measurements (for more details see above, 7.4.3):

i) Demographics ii) Upper Airway iii) Blood tests iv) Symptom and Quality of Life scores v) NIV usage

Patients will be given a debriefing by the study team and individual study reports can be requested at this stage, they will be provided once the entire analysis has been completed.

Definition of End of Trial

The trial finishes with the 12-week follow up assessment. The patients will then be referred back to standard care to be followed up in the outpatient setting at the Lane Fox Unit.

ELIGIBILITY:
Inclusion Criteria:

* hypercapnic respiratory failure (PaCO2 > 6kPa)
* low usage of home mechanical ventilation (NIV < 4hours/night).
* body mass index (BMI) >18.5kg/m2
* all genders
* age 18-90years.

Exclusion Criteria:

* no hypercapnic respiratory failure (PaCO2<6kPa)
* no sleep-disordered breathing (AHI<5/hour)
* exclusively obstructive sleep apnoea
* isolated Rapid-Eye-Movement (REM) sleep associated OSA
* cachexia (BMI <18.5 kg/m2)
* severe pulmonary hypertension
* valvular heart disease
* heart failure (New York Heart Association, NYHA III-IV)
* myocardial infarction and significant cardiac arrhythmias
* uncontrolled hypertension
* active psychiatric disease
* co-existing non-respiratory sleep disorder.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Adherence | 3 months
  Usage / night (hours)

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | 3 months
  0-24 points (higher results indicate increased levels of sleepiness)
Stanford Sleepiness Scale | 3 months
  0-7 points (higher scores indicate more symptoms)
Hospital Anxiety and Depression Scale | 3 months
  0-42 points (higher scores indicate more symptoms)
Severe Respiratory Insufficiency Questionnaire | 3 months
  points (higher scores indicate more symptoms)
EQ-5D | 3 months
  0-100 points (higher scores indicate better functioning and quality of life)
Healthcare Resource Usage | 3 months
  contacts with GP/hospital
Arterial Blood Gas analysis | 3 months
  kPA
SpO2 | 3 months
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon request data can be shared according to ethics committee and national guidelines and laws, as well as GDPR requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within one year following completion of the trial
Access Criteria: upon request

REFERENCES:
- [Derived] Alsharifi A, Kaltsakas G, Ramsay M, Owusu-Afriyie J, Radcliffe G, Rafferty G, Steier J. Remote monitoring to improve low adherence in non-invasive ventilation: a protocol for a randomised controlled clinical trial (READ-NIV trial). J Thorac Dis. 2024 Sep 30;16(9):6263-6271. doi: 10.21037/jtd-24-86. Epub 2024 Sep 4. PMID 39444901